CLINICAL TRIAL: NCT00493454
Title: Multicenter Phase II Study for Zevalin® in Patients With Relapsed/Refractory Indolent Lymphomas: Extranodal Marginal Lymphoma of MALT Type, Nodal Marginal Zone B-Cell Lymphoma, and Splenic Marginal B-Cell Lymphoma
Brief Title: Ibritumomab Tiuxetan for Treatment of Non-Follicular CD20+ Indolent Lymphomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0571
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Lymphoma
Keywords: Indolent Lymphoma; Extranodal Marginal; Nodal Marginal Zone; Splenic Marginal; MALT Type; Zevalin; Ibritumomab Tiuxetan; Rituximab
MeSH Terms: conditions — Lymphoma | interventions — ibritumomab tiuxetan; Rituximab; Indium-111

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibritumomab tiuxetan + Rituximab (Experimental): Rituximab 250 mg/m² intravenous (IV) Days 1 and 8, 111In Ibritumomab Tiuxetan (5mCi of 111In, 1.6 mg of Ibritumomab Tiuxetan) IV (over 10 minutes) on Day 1; and 90Y Ibritumomab Tiuxetan 0.3 or 0.4 mCi/kg IV (over 10 minutes) on Day 8 after the Day 8 of Rituximab.
  Interventions: Drug: Zevalin; Drug: Rituximab; Drug: ^111 In Ibritumomab Tiuxetan

INTERVENTIONS:
Drug: Zevalin — .3 mCi IV Over 10 Minutes x 1 Day
  Other Names: Ibritumomab Tiuxetan
Drug: Rituximab — 250 mg/m^2 IV Over 6 to 8 Hours
Drug: ^111 In Ibritumomab Tiuxetan — 1.6 mg IV Over 10 Minutes x 1 Day
  Other Names: Indium-111

SUMMARY:
Primary Objective:

* Overall Response Rate (ORR).

Secondary Objectives:

* The Duration of Response (DR) and Time to Treatment Progression (TTP) in all patients and in the responders.
* Complete Responses (CR)/Complete Responses unconfirmed (CRu), and Partial Responses (PR).
* Time to next anticancer therapy (TTNT).

DETAILED DESCRIPTION:
^90 Y Ibritumomab tiuxetan and rituximab are both designed to attach to lymphoma cells, causing them to die.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a physical exam. Your blood (about 2 to 3 teaspoons) and urine will be collected for routine tests. You will have a chest x-ray and computerized tomography (CT) scans of the neck, chest, abdomen, and pelvis. You will have a bone marrow aspirate and biopsy performed. To collect a bone marrow aspirate and biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. Women who are able to have children must have a negative blood pregnancy test.

The study doctors will first make sure that your disease has not spread too much and is not too severe to require immediate treatment with chemotherapy before you can begin treatment on this study. If you are found to be eligible to take part in this study, you will be given Benadryl (diphenhydramine) by vein, and you will be given Tylenol (acetaminophen) by mouth before each dose of rituximab. This is done to help decrease the risk of developing side effects of rituximab. You will then receive 1 dose of rituximab by vein over 6 to 8 hours on Day 1 of treatment. After treatment with rituximab, you will then be given a radioactive antibody, ^111 In Ibritumomab tiuxetan (this is a radioactive agent that binds to rituximab to help with imaging exams), by vein over about 10 minutes. This is so researchers can use a special camera to see where the drug is in your body.

You will have imaging performed (with the special camera) on Day 1 and on either Day 2 or Day 3. On Day 8, you will receive a second dose of rituximab. This will then be followed by a dose ^90 Y Ibritumomab tiuxetan of given by vein over 10 minutes. This completes the treatment.

If you experience intolerable side effects while on this study, you may be removed from this study. The study doctor will then offer other treatment options to you.

For your follow-up, you will have blood (about 2 tablespoons) drawn once a week for the first 3 months, then every 3 months for 1 year, and then every 4 months for the second year. At these visits, you may also have CT scans, x-rays, and bone marrow biopsies and aspirates performed, if needed.

This is an investigational study. ^90 Y Ibritumomab tiuxetan and rituximab have been approved by the FDA for the treatment of indolent B-cell lymphoma. Up to 35 patients will take part in this multicenter study. Up to 15 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. No anti-cancer therapy for three weeks (six weeks if Rituximab, nitrosourea or Mitomycin C) prior to study initiation, and fully recovered from acute toxicities associated with prior surgery, radiation treatments, chemotherapy, or immunotherapy.
2. Previously treated patients with a histology of refractory/relapsed indolent lymphomas including: (a) Extranodal marginal lymphoma of MALT type; (b) Nodal Marginal zone B-cell lymphoma (+/- monocytoid cells); (c) Splenic marginal B-cell lymphoma (+/- villous lymphocytes).
3. Signed informed consent
4. Age >/= 18 years
5. Expected survival >/= 3 months
6. Pre-study Zubrod performance status of 0, 1, or 2
7. Acceptable hematologic status within two weeks prior to patient registration, including: (a) Absolute neutrophil count ([segmented neutrophils + bands] * total white blood count (WBC)) >/= 1,500/mm^3; (b) Platelet counts >/= 100,000/mm^3.
8. Female patients who are not pregnant or lactating
9. Men and women of reproductive potential who are following accepted birth control methods (as determined by the treating physician)
10. Patients previously on Phase II drugs if no long-term toxicity is expected, and the patient has been off the drug for eight or more weeks with no significant post treatment toxicities observed
11. Patients determined to have < 25% bone marrow involvement with lymphoma within six weeks of registration (define measurement of a bone marrow aspirate or biopsy) (This criteria must be strictly met for adequate patient safety.)
12. Patient should have at least one lesion measuring >/= 2 cm in a single dimension.

Exclusion Criteria:

1. Prior myeloablative therapies with autologous bone marrow transplantation (ABMT) or peripheral blood stem cell (PBSC) rescue.
2. Platelet count< 100,000 cells/mm^3.
3. Presence of hypocellular bone marrow.
4. Patients with history of failed stem cell collection.
5. Prior radioimmunotherapy
6. Presence of Central Nervous System (CNS) lymphoma
7. Patients with HIV.
8. Patients with pleural effusion
9. Patients with abnormal liver function: total bilirubin > 2.0 mg/dL
10. Patients with abnormal renal function: serum creatinine > 2.0 mg/dL
11. Patients who have received prior external beam radiation therapy to > 25% of active bone marrow (involved field or regional)
12. Patients who have received short-acting growth factor support (Leukine, Neupogen, Procrit) within 2 weeks prior to treatment or long-acting growth-factor support (Aranesp), Neulasta) within 4 weeks prior to treatment.
13. Serious nonmalignant disease or infection which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives
14. Major surgery, other than diagnostic surgery, within four weeks
15. Evidence of transformation in the latest biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Samaniego, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center Official Web Site — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 13, 2006 to November 8, 2007. All participants recruited in medical clinic at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Ibritumomab Tiuxetan + Rituximab
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ibritumomab Tiuxetan + Rituximab
Number analyzed (Participants) | 6
Age Continuous [Median (Full Range); unit: years] | 67.5 [55 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate (ORR) = number of participants out of all participating with Complete Response (CR) + Partial Response (PR) as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Partial response (PR) must have ≥ 30% decrease in the sum of longest diameter of all target lesions, from the baseline sum. Complete response (CR) must have disappearance of all target and non-target lesions. Response assessed by magnetic resonance imaging (MRI) or computed tomography (CT) scans, every 3 months for the first year and every 6 months up to 3 years following.
Time Frame: Evaluation 4 weeks after administration of Zevalin up to 3 years
Population: One participant did not receive treatment and was excluded from analysis.
Measure: Number; unit: proportion of participants
Arm/Group | Ibritumomab Tiuxetan + Rituximab
Number analyzed (Participants) | 5
proportion of participants | 0.8

ADVERSE EVENTS:
Time Frame: 4 years and 4 months
Arm/Group | Ibritumomab Tiuxetan + Rituximab
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibritumomab Tiuxetan + Rituximab (N=5)
Neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibritumomab Tiuxetan + Rituximab (N=5)
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No